CLINICAL TRIAL: NCT06819800
Title: The Effect of Three Different Nasogastric Tube Fixation Materials on Pressure Injury in the Intensive Care Unit
Brief Title: The Effect of Three Different Nasogastric Tube Fixation Materials on Pressure Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ayse_kaya_61
Record Dates: First submitted 2025-01-08; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pressure Ulcer; Nursing Care
Keywords: Intensive Care Unit; nasogastric tube fixation; pressure injury; medical equipment; nursing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The study was conducted with 3 groups. The experimental groups consisted of medical silk plaster and transparent waterproof plaster groups. The control group consisted of the elastic bandage group, which was routinely applied in intensive care unit. Patients were randomly assigned to the groups and 3 different fixation materials were applied according to their group. Fixation materials were changed every 24 hours and skin care was performed. Patients were followed up until discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic Flaster (Active Comparator): Elastic Flaster:
  Elastic flaster is a hypoallergenic therapeutic product and is made of an elastic, non-woven fabric. It has a polyacrylate adhesive, which allows it to be easily fixed. Thanks to its porous structure, it allows air intake, recognition and moisture permeability. Elastic plasters, which easily adapt to the connections with their flexible structure body structures, adapt to the natural movements of the skin and increase the comfort of the patient. This feature may be especially preferred for patients who move a lot. Although elastic dressings are generally more affordable than other types of dressings, they may increase costs in the long term due to frequent replacement. In the Intensive Care Unit, elastic plasters are routinely used for nasogastric tube fixation.
  Interventions: Other: Elastic Flaster
- Medical Silk Flaster (Experimental): Medical Silk Flasters:
  Medical silk flaster is a medical material made of acetate silk with rubber-based fittings containing mineral oxide. It is used for fixation in surgical applications. It is effective in fixing materials such as catheters, cover cloths and wound dressings thanks to its strong adhesive properties. The material used in its content provides a clean appearance compatible with the skin and increases comfort. However, this type of flasters may cause skin irritation in some patients with prolonged use. The cost of silk flasters is moderate, and their high adhesive properties make them cost-effective in the long term as they require fewer changes.
  Interventions: Other: Medical Silk Flaster
- Transparent Waterproof Flaster (Experimental): Transparent Waterproof Waterproof Flaster The transparent waterproof patch is a hypoallergenic product suitable for sensitive skin. It offers an ideal use for the storage of maintenance and repair areas. It is effectively used for fixing the number of medical supplies. The transparent structure allows for clearer observation of operations. These flasters perform well even in humid environments and reduce the risk of infection. It has a strong adhesive, long-lasting feature and does not cause any residue on the skin after use. It can be easily torn by hand both transversely and longitudinally, ensuring user practicality.
  Interventions: Other: Transparent Waterproof Flaster

INTERVENTIONS:
Other: Transparent Waterproof Flaster — Patients determined by randomization method were divided into three groups. "Patient Information Form", 'Patient Follow-up Form', 'Glasgow Coma Scale' and 'Braden Pressure Ulcer Risk Assessment Scale' were applied to the patients in the transparent waterproof flaster group, one of the experimental groups. Nasogastric tube care was applied at 24-hour intervals. The dorsum of the nose was first cleaned with saline and then disinfected with a skin antiseptic containing alcohol and chlorhexidine gluconate. Afterwards, a transparent waterproof flaster was applied. The transparent waterproof flaster was prepared using the "nasal preparation by pants tape method" technique. Afterwards, the "Patient Follow-up Form", "Glasgow Coma Scale" and "Braden Pressure Injury Risk Diagnostic Scale" were re-administered by the investigator at 72 hours and at discharge. If pressure injury developed, the "Nasogastric Tube-Related Pressure Injury Staging Form" was completed.
  Arms: Transparent Waterproof Flaster
Other: Medical Silk Flaster — Patients determined by randomization method were divided into three groups. "Patient Information Form", 'Patient Follow-up Form', 'Glasgow Coma Scale' and 'Braden Pressure Wound Risk Assessment Scale' were applied to the patients in the medical silk flaster group, one of the experimental groups. Nasogastric tube care was applied at 24-hour intervals. The dorsum of the nose was first cleaned with saline and then disinfected with a skin antiseptic containing alcohol and chlorhexidine gluconate. Afterwards, a medical silk flaster was applied. The medical silk flaster was prepared using the "nasal preparation by pants tape method" technique. Afterwards, the "Patient Follow-up Form", "Glasgow Coma Scale" and "Braden Pressure Injury Risk Diagnostic Scale" were re-administered by the investigator at 72 hours and at discharge. If pressure injury developed, the "Nasogastric Tube-Related Pressure Injury Staging Form" was completed.
  Arms: Medical Silk Flaster
Other: Elastic Flaster — Patients determined by randomization method were divided into three groups. "Patient Information Form", 'Patient Follow-up Form', 'Glasgow Coma Scale' and 'Braden Pressure Wound Risk Assessment Scale' were administered to the patients in the control group, which was in the elastic flaster group. Nasogastric tube care was applied at 24-hour intervals. The dorsum of the nose was first cleaned with saline and then disinfected with a skin antiseptic containing alcohol and chlorhexidine gluconate. Afterwards, an elastic flaster was applied. The elastic flaster was prepared using the "preparation of the nose by the pants tape method" technique. Afterwards, the "Patient Follow-up Form", "Glasgow Coma Scale" and "Braden Pressure Injury Risk Diagnostic Scale" were re-administered by the investigator at 72 hours and at discharge. If pressure injury developed, the "Nasogastric Tube-Related Pressure Injury Staging Form" was completed.
  Arms: Elastic Flaster

SUMMARY:
This randomized controlled experimental study aims to comparatively determine the effects of three different nasogastric tube fixation materials (elastic plaster, medical silk plaster, transparent waterproof plaster) on pressure injuries in adult patients hospitalized in ICU.

This study was carried out in the Intensive Care Units (ICU) of a university-affiliated training and research hospital in Istanbul, Turkey. 84 patients were divided into three groups of 28 patients each, and were fixed with different materials. Data were collected using the Patient Information Form, Patient Follow-up Form, Braden Pressure Wound Risk Assessment Scale, Glasgow Coma Scale, and Nasogastric Tube-Related Pressure Injuries Staging and Follow-up Form. The data were analyzed using the Statistical Package for Social Sciences (SPSS) v27 statistical analysis program. The frequency and severity of pressure injuries between groups were evaluated by statistical methods such as Chi-square analysis, analysis of variance and Bonferroni test.

DETAILED DESCRIPTION:
Purpose and Design Type of the Study The aim of this study with a randomized controlled experimental design was to examine the effects of three different nasogastric tube fixation materials on pressure injury in adult patients hospitalized in the Intensive Care Unit (ICU).

Research Hypothesis H0: Different nasogastric tube fixation materials have no significant effect in preventing pressure injuries.

H1: Different nasogastric tube fixation materials have a significant effect on preventing pressure injuries.

Variables of the Study Dependent Variables: Pressure injury development. Independent Variables: Three different nasogastric tube fixation materials and individual/disease characteristics of patients.

Place and Time of the Study This study was conducted between December 28, 2023 and June 2024 in the Intensive Care Units (ICU) of a university-affiliated training and research hospital in Istanbul.

Study Population and Sample The population of the study consisted of adult patients undergoing inpatient care and treatment in the intensive care units of a university-affiliated training and research hospital in Istanbul, who were administered nasogastric tubes. The sample was determined as a minimum of 84 patients (n1=28, n2=28, n3=28) using G*Power 3.0.10 software with 90% power, 5% margin of error and f=0.20 effect size. The material group to which the patients were assigned was determined by randomization. In this context, the randomization table was created using an online platform (https://www.random.org/sequences/?min=1&max =84&col=3&format=html&rnd=new). The first column was considered as the first experimental group (medical silk plaster), the second column as the second control group (transparent waterproof plaster), and the third column as the control group (elastic plaster). Due to the nature of the study, blinding could not be performed because the researcher and the participant were aware of the intervention.

Inclusion and exclusion criteria Patients to be included in the study;

* Between the ages of 18-65
* Duration of hospitalization in the ICU should be at least 24 hours
* Having no cognitive and affective problems
* Nasogastric (NG) tube insertion for the first time and tube placement for at least 72 hours
* Nasogastric tube maintenance at least once a day
* Glasgow Coma Scale (GCS) score of 9 and above
* Oxygen support is not provided with medical devices
* No skin problem that may prevent skin diagnostics
* No burns/trauma/operation on the face and nose area
* No history of pressure injury to the nose
* Not having a diagnosis of diabetes mellitus (DM). Exclusion criteria;
* Under 18 or over 65 years of age
* Having a state of consciousness or affective problem(s)
* GCS score below 9
* The presence of facial problem(s) that may prevent nasogastric tube administration.

Data Collection Tools Patient information questionnaire The information form developed to evaluate the socio-demographic and disease characteristics of the patients was prepared by the investigators under the guidance of the relevant literature. The form consists of two parts and includes the socio-demographic data of the patients after the nasogastric tube was applied for the first time. The form was administered to the patients on the first day to collect these data.

Patient follow-up questionnaire This form, which was created according to the shift hours of the nurses, was prepared by the researchers based on the relevant literature in order to record the patients' vital signs, laboratory values and diagnoses related to the nasal region. This form was administered to patients who met the sampling criteria on the day of nasogastric tube insertion, at 72 hours and at discharge.

Glasgow coma scale (GCS) The GCS, developed in 1974 in Glasgow, Scotland, is a common scale used to assess the state of consciousness of comatose patients. It consists of three parameters, namely "eye clarity", "verbal and motor response". The total score ranges from 3 to 15, with 3 points indicating deep coma and 15 points indicating full awareness and alertness. It was administered by the investigator to patients who met the sampling criteria on the day of nasogastric tube insertion, at 72 hours and at discharge. In this study, the cronbach alpha value was 0.726 on the first day, 0.839 on the third day, and 0.894 on the last day. Braden pressure sore risk assessment scale Developed in 1984 by Braden and used to assess pressure sore risk factors, this scale was improved by Braden and Bergstrom in 1987. The subscales of the scale include stimulus perception, activity, movement, moisture, nutrition and friction-tearing. The scores obtained from the subscales constitute the total scale score. The score range is 6-23, and the lower the score, the higher the risk of developing pressure sores. According to the scale score, risk levels are classified as "12 and below high risk", "13-14 medium risk", "15-16 low risk". In people aged 75 years and older, a score of 15-18 is considered low risk. The first reliability study of the scale in Turkey was conducted in 1997 and the reliability coefficient was found to be 0.95. In this study, cronbach's alpha value was 0.610 on the first day, 0.632 on the third day, and 0.639 on the last day.

Nasogastric tube-related pressure injuries follow-up questionnaire This form was developed to stage and monitor pressure injuries and was based on the classification guidelines developed by EPUAP and NPUAP. In this study, this form was applied by the researcher to patients with pressure injury.

Medical Tools and Equipment Used in the Data Collection Phase Materials to be used in nasogastric tube fixation and their properties Within the scope of the study, three different materials, elastic, medical silk and transparent waterproof plaster, were applied to provide fixation in patients who underwent nasogastric tube placement. In the application, which plaster to be used in the patients was determined by the researchers by randomization Elastic plaster It is a hypoallergenic treatment product and is made of an elastic non-woven fabric. It has a polyacrylate adhesive, which makes it easy to fix. Thanks to its porous structure, it allows airing, recognition and moisture permeability. Elastic bandages, which easily adapt to the connections with their flexible structure body structures, adapt to the natural movements of the skin and increase the comfort of the patient. This feature is especially preferable for patients who move a lot. Although elastic dressings are generally more affordable than other types of dressings, they can increase costs in the long term due to frequent replacement. In the Intensive Care Unit, elastic packing is routinely used for nasogastric tube fixation.

Medical silk plaster It is a medical material made of acetate silk with rubber-based fittings containing mineral oxide. It is used for fixation in surgical applications. It is effective in the fixation of materials such as catheters, cover cloths and wound dressings thanks to its strong adhesive properties. The material used in its content provides a clean appearance compatible with the skin and increases comfort. However, this type of plasters may cause skin irritation in some patients with prolonged use. The cost of silk plasters is moderate, and their high adhesive properties make them cost-effective in the long run, as they require fewer changes.

Transparent waterproof plaster It is a hypoallergenic product suitable for sensitive skin. It is ideal for storing maintenance and repair areas. It is used effectively in fixing the number of medical supplies. Thanks to the transparent structure, it provides clearer observation of the procedures. These plasters perform well even in humid environments and reduce the risk of infection. It has a strong adhesive, long-lasting feature and does not cause any residue on the skin after use. It can be easily torn both transversely and longitudinally by hand and the user's practicality is ensured. Research Implementation Before the research data were collected, ethical approval (20.09.2022-78405) was obtained from the non-interventional clinical research ethics committee of a foundation university and institutional permission (19.12.2023-2023/20) was obtained from a university-affiliated training and research hospital in Istanbul. After the necessary permissions were approved, the investigators identified the patients who had nasogastric tube insertion and met the sampling criteria, informed them and obtained written informed consent. Which fixation material would be applied to the patients was determined by randomization method and the patients were divided into three groups. Then, "Patient Information Questionnaire", "Patient Follow-up Questionnaire", "Glasgow Coma Scale" and "Braden Pressure Ulcer Risk Assessment Scale" were administered to the patients with nasogastric tube insertion in the order in the research design scheme. The investigator administered nasogastric tube care to each patient who met the sampling criteria at 24-hour intervals in accordance with the standard protocol in the intensive care unit. During this care process, the back of the patient's nose was first cleaned with saline and then disinfected with a skin antiseptic containing alcohol and chlorhexidine gluconate. Afterwards, the fixation material determined by randomization method was carefully prepared for each patient. According to the standard protocol of the Intensive Care Unit, the fixation of the nasogastric tube, which was performed only by the investigator, was performed in a single session using three different materials. The three different fixation materials were prepared using the "nasal preparation by pants tape method" technique described below. Each fixation material was cut 10 cm in length and 2.5 cm in width and cut in half. The uncut part of the prepared material was fixed to the nasal dorsum, while the halved ends were wrapped around the nasogastric tube in opposite directions to complete the fixation process. All these procedures were performed using a sterile technique and observing the vital parameters of the patient. This procedure was performed separately by the investigator for each patient using three different fixation materials according to the same protocols. Afterwards, the "Patient Follow-up Form", "Glasgow Coma Scale" and "Braden Pressure Injury Risk Diagnostic Scale" were re-administered to the patient by the investigator at 72 hours and during discharge. When pressure injury developed, the "Nasogastric Tube-Related Pressure Injury Follow-up Questionnaire" was completed and the stage and extent of the pressure injury were recorded and reported in detail.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Duration of hospitalization in the ICU should be at least 24 hours
* Having no cognitive and affective problems
* Nasogastric (NG) tube insertion for the first time and tube placement for at least 72 hours
* Nasogastric tube maintenance at least once a day
* Glasgow Coma Scale (GCS) score of 9 and above
* Oxygen support is not provided with medical devices
* No skin problem that may prevent skin diagnostics
* No burns/trauma in the face and nose area/operation not to spend
* No history of pressure injury to the nose
* The absence of a diagnosis of Diabetes Mellitus (DM) was determined.

Exclusion Criteria:

* Under 18 or over 65 years of age
* Having a state of consciousness or affective problem(s)
* GCS score below 9
* The presence of facial problem(s) that may prevent nasogastric tube insertion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale | Baseline, 72 hours and average 15 days
  Developed in Glasgow, Scotland in 1974, the GCS is a common scale used to assess the state of consciousness of comatose patients. It consists of three parameters: "eye openness", "verbal and motor response". The total score ranges from 3 to 15, with 3 points indicating deep coma and 15 points indicating full awareness and alertness.
Braden Pressure Ulcer Risk Assessment Scale | Baseline, 72 hours and average 15 days
  Developed in 1984 by Braden and used to assess pressure sore risk factors, this scale was improved by Braden and Bergstrom in 1987. The subscales of the scale include stimulus perception, activity, movement, moisture, nutrition and friction-tearing. The scores obtained from the sub-dimensions constitute the total scale score. The score range is 6-23, and the lower the score, the higher the risk of developing pressure sores. According to the scale score, risk levels are classified as "12 and below high risk", "13-14 medium risk", "15-16 low risk". A score of 15-18 is considered low risk in people aged 75 years and older.

SECONDARY OUTCOMES:
Nasogastric Tube Related Pressure Injuries Follow-up Questionnaire | on average 10-15 days after the wound is formed in the patient
  This form is used for staging and monitoring pressure injuries.
patient information questionnaire | Baseline
  The information questionnaire, which was developed to evaluate the socio-demographic and disease characteristics of the patients, was prepared by the investigators under the guidance of the relevant literature. The questionnaire consisted of two parts and included the socio-demographic data of the patients after the nasogastric tube was applied for the first time. The questionnaire was administered to the patients on the first day to collect these data.
patient nasal area monitoring questionnaire | Baseline, 72 hours and average 15 days
  This questionnaire, which was created according to the shift hours of the nurses, was prepared by the researchers based on the relevant literature in order to record the patients' vital signs, laboratory values and diagnoses related to the nasal region. This questionnaire was administered to patients who met the joint criteria on the day of nasogastric tube insertion, at 72 hours and on average 15 days.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakıf University, Istanbul, Eyüp Sultan
  - Bezmialem Vakif University, Istanbul, Eyüpsultan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [2] Karadağ A, Karabağ AA. (2013)Basınç Ülserlerinde Etiyoloji ve Fizyopatoloji. Baktıroğlu S, Aktaş Ş editörler. Kronik Yarada Güncel Yaklaşımlar, 1. Baskı. İstanbul.116-209
- [Background] Neill S, Martin D. Nursing care bundles in the prevention of medical device related pressure ulcers: An integrative review. J Tissue Viability. 2024 Aug;33(3):376-386. doi: 10.1016/j.jtv.2024.04.003. Epub 2024 Apr 10. PMID 38641481
- [Background] Coyer FM, Stotts NA, Blackman VS. A prospective window into medical device-related pressure ulcers in intensive care. Int Wound J. 2014 Dec;11(6):656-64. doi: 10.1111/iwj.12026. Epub 2013 Feb 4. PMID 23374630
- [Background] Apold J, Rydrych D. Preventing device-related pressure ulcers: using data to guide statewide change. J Nurs Care Qual. 2012 Jan-Mar;27(1):28-34. doi: 10.1097/NCQ.0b013e31822b1fd9. PMID 21826028
- [Background] [6] Black JM, Kalowes P.(2016) Medical device-related pressure ulcers. Chronic Wound Care Management and Research.3:91- 99.
- [Background] [7] Çelik, N. (2013). Nazogastrik tüp ve hemşirelik girişimleri. SD Ü Sağlık Bilimleri Enstitüsü Dergisi, 4(2), 108-113.
- [Background] Tayyib N, Asiri MY, Danic S, Sahi SL, Lasafin J, Generale LF, Malubay A, Viloria P, Palmere MG, Parbo AR, Aguilar KE, Licuanan PM, Reyes M. The Effectiveness of the SKINCARE Bundle in Preventing Medical-Device Related Pressure Injuries in Critical Care Units: A Clinical Trial. Adv Skin Wound Care. 2021 Feb 1;34(2):75-80. doi: 10.1097/01.ASW.0000725184.13678.80. PMID 33443912
- [Background] [9] Holomuzki, M., DeVilliers, A. ve Kuhn, M. (2017). *ÖnlemekNazogastrik tüp HAPU'larının önlenmesi . Ulusalhttps://www.nacns.org/wp -content /uploads /2017 /03 /Poster-
- [Background] Kisting MA, Korcal L, Schutte DL. Lose the Whoosh: An Evidence-Based Project to Improve NG Tube Placement Verification in Infants and Children in the Hospital Setting. J Pediatr Nurs. 2019 May-Jun;46:1-5. doi: 10.1016/j.pedn.2019.01.011. Epub 2019 Feb 21. PMID 30798144
- [Background] Yuksel A, Ugur KS, Kizilbulut G, Ark N, Kurtaran H, Kaya M, Gunduz M. Long-term results of one staged multilevel surgery with tongue suspension surgery or one level palatal surgery for treatment of moderate and severe obstructive sleep apnea. Eur Arch Otorhinolaryngol. 2016 May;273(5):1227-34. doi: 10.1007/s00405-015-3813-4. Epub 2016 Jan 29. PMID 26825802
- [Background] [12] Nursing Management of Nasogastric Tube Feeding in Adult Patients, Moh Nursing Clinical Practice Guidelines 1/2010.
- [Background] [13] Sivrikaya, S., & Sarıkaya, S.(2020) Yoğun Bakım Hastalarında Bası Ülseri, Önleme Ve Hemşirelik Bakımı. Yoğun Bakım Hemşireliği Dergisi , 24 (2), 139-149.
- [Background] [14] Tezcan, B., & Karabacak, B. G. (2021). Basınç Yaralanmalarının Önlenmesinde Daha İyi Sonuçlara Doğru: Kanıta Dayalı Uygulamalar. Balıkesir Sağlık Bilimleri Dergisi, 10(1), 49-54.
- [Background] [15] Reith, F., Van den Brande, R., Synnot, A., Gruen, R., & Maas, AI (2016). Glasgow Koma Ölçeğinin güvenilirliği: sistematik bir inceleme. Yoğun bakım tıbbı , 42 (1), 3-15.
- [Background] Ayello EA, Braden B. How and why to do pressure ulcer risk assessment. Adv Skin Wound Care. 2002 May-Jun;15(3):125-31; quiz 132-33. doi: 10.1097/00129334-200205000-00008. PMID 12055446
- [Background] Bergstrom N, Braden B, Kemp M, Champagne M, Ruby E. Predicting pressure ulcer risk: a multisite study of the predictive validity of the Braden Scale. Nurs Res. 1998 Sep-Oct;47(5):261-9. doi: 10.1097/00006199-199809000-00005. PMID 9766454
- [Background] Bergstrom N, Braden BJ, Laguzza A, Holman V. The Braden Scale for Predicting Pressure Sore Risk. Nurs Res. 1987 Jul-Aug;36(4):205-10. PMID 3299278
- [Background] Zeng LA, Lie SA, Chong SY. Comparison of Medical Adhesive Tapes in Patients at Risk of Facial Skin Trauma under Anesthesia. Anesthesiol Res Pract. 2016;2016:4878246. doi: 10.1155/2016/4878246. Epub 2016 Jun 12. PMID 27382368
- [Background] McNichol L, Lund C, Rosen T, Gray M. Medical adhesives and patient safety: state of the science: consensus statements for the assessment, prevention, and treatment of adhesive-related skin injuries. Orthop Nurs. 2013 Sep-Oct;32(5):267-81. doi: 10.1097/NOR.0b013e3182a39caf. PMID 24022422
- [Background] Hinrichs-Krapels S, Ditewig B, Boulding H, Chalkidou A, Erskine J, Shokraneh F. Purchasing high-cost medical devices and equipment in hospitals: a systematic review. BMJ Open. 2022 Sep 1;12(9):e057516. doi: 10.1136/bmjopen-2021-057516. PMID 36581959
- [Result] [1] EUAP-PPPIA (European Pressure Ulcer Advisory Panel- National Pressure Ulcer Advisory PanelPan Pacific Pressure Injury Alliance) 2014. Prevention and Treatment of Pressure ulcers: Quick reference guide. ISBN-13: 978-0-9579343-6-https://www.epuap.org/wp content/uploads/2010/10/NPUAP-EPUAPPPPIA-Quick-Reference-Guide-2014-DIGITAL.pdf.